CLINICAL TRIAL: NCT01862926
Title: A Randomized, Double Blind Controlled Trial Comparing Rituximab Against Intravenous Cyclophosphamide in Connective Tissue Disease Associated Interstitial Lung Disease
Brief Title: Rituximab Versus Cyclophosphamide in Connective Tissue Disease-ILD
Acronym: RECITAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); University of East Anglia (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBHIPF004; 2012-003633-42 (EudraCT Number)
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Interstitial Lung Disease; Scleroderma; Idiopathic Inflammatory Myositis; Mixed Connective Tissue Disease
Keywords: connective tissue disease; interstitial lung disease; pulmonary fibrosis; rituximab; scleroderma; polymyositis; dermatomyositis
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Diffuse; Myositis; Mixed Connective Tissue Disease; Connective Tissue Diseases; Pulmonary Fibrosis; Polymyositis; Dermatomyositis | interventions — Rituximab; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): 1g given at baseline and two weeks.
  Interventions: Drug: Rituximab
- Cyclophosphamide (Active Comparator): Intravenous dose of 600 mg/m2 body surface area. 6 doses given 4 weekly.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Rituximab
  Arms: Rituximab
Drug: Cyclophosphamide
  Arms: Cyclophosphamide

SUMMARY:
Interstitial lung disease (ILD) is characterised by inflammation and scarring of the lung and is the leading cause of death in patients with systemic sclerosis, and contributes significantly to morbidity and mortality in many other connective tissue diseases (CTDs) such as polymyositis/dermatomyositis and mixed connective tissue disease. When ILD is extensive and/or progressive, immunosuppressive medication is often required to stabilize lung disease and alleviate symptoms. Current standard care for CTD associated ILD is extrapolated from studies performed in individuals with systemic sclerosis and comprises low dose corticosteroids and intravenous cyclophosphamide followed by oral azathioprine. In some individuals even this intensive immunosuppression is insufficient to prevent deterioration, and in a significant minority of affected individuals this results in respiratory failure and death. Rituximab has recently been reported as an effective 'rescue therapy' for stabilizing and even improving ILD in this patient group. Based on observations gained from this experience, the investigators believe that rituximab is a potential important alternative to current best therapy for this patient group. This study has therefore been initiated to evaluate the efficacy of rituximab (compared with standard therapy) in patients with progressive CTD related ILD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years at visit 1
* A diagnosis of connective tissue disease, based on internationally accepted criteria, in one of the following categories21-24: (see Appendix 1 for details)

  * Systemic sclerosis
  * Idiopathic interstitial myopathy (including polymyositis/dermatomyositis)
  * Mixed connective tissue disease
* Severe and/or progressive interstitial lung disease associated with the underlying connective tissue disease.
* Chest HRCT performed within 12 months of study visit 1
* Intention of the caring physician to treat the ILD with intravenous cyclophosphamide (with treatment indications including deteriorating symptoms attributable to ILD, deteriorating lung function tests, worsening gas exchange or extent of ILD at first presentation) and where there is a reasonable expectation that immunosuppressive treatment with stabilize or improve CTD-ILD. In individuals with scleroderma it is anticipated that subjects will fulfil the criteria for extensive disease defined by Goh et al19
* Able to provide written informed consent

Exclusion Criteria:

* Age <18 or >80 years.
* Previous treatment with rituximab and/or intravenous cyclophosphamide
* Known hypersensitivity to rituximab or cyclophosphamide or their components
* Significant (in the opinion of the investigator) other organ co-morbidity including cardiac, hepatic or renal impairment
* Co-existent obstructive pulmonary disease (e.g. asthma, COPD, emphysema) with pre bronchodilator FEV1/FVC < 70%
* Patients at significant risk for infectious complications following immunosuppression, including; HIV positive or other immunodeficiency syndromes (including hypogammaglobulineamia)
* Suspected or proven untreated tuberculosis
* Viral hepatitis
* Infection requiring antibiotic treatment in the preceding four weeks
* Unexplained neurological symptoms (which may be suggestive of progressive mutifocal leukoencephalopathy; PML). Neurological symptoms arising as a consequence of the underlying CTD do not necessitate exclusion.
* Other investigational therapy (participation in research trial) received within 8 weeks of visit 1
* Immunosuppressive therapy (other than corticosteroids) received within 2 weeks of visit 1 (randomization)
* Pregnant or breast feeding women, or women of child-bearing potential, not using a reliable contraceptive method
* Unexplained haematuria, or previous bladder carcinoma
* Unable to provide informed written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Absolute change in FVC | 48 weeks

SECONDARY OUTCOMES:
• Change from baseline in diffusing capacity for carbon monoxide (DLco) | 48 weeks
• Change from baseline in health related quality of life scores | 48 weeks
• Change from baseline in global disease activity score | 48 weeks
• Progression free survival | 48 weeks
  composite endpoint of mortality, transplant, treatment failure or decline in FVC > 10% compared to baseline
• Adverse and serious adverse events (as defined in GCP) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toby M Maher, MD PhD, Study Chair — Royal Brompton and Harefield Foundation NHS Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Background] Tyndall AJ, Bannert B, Vonk M, Airo P, Cozzi F, Carreira PE, Bancel DF, Allanore Y, Muller-Ladner U, Distler O, Iannone F, Pellerito R, Pileckyte M, Miniati I, Ananieva L, Gurman AB, Damjanov N, Mueller A, Valentini G, Riemekasten G, Tikly M, Hummers L, Henriques MJ, Caramaschi P, Scheja A, Rozman B, Ton E, Kumanovics G, Coleiro B, Feierl E, Szucs G, Von Muhlen CA, Riccieri V, Novak S, Chizzolini C, Kotulska A, Denton C, Coelho PC, Kotter I, Simsek I, de la Pena Lefebvre PG, Hachulla E, Seibold JR, Rednic S, Stork J, Morovic-Vergles J, Walker UA. Causes and risk factors for death in systemic sclerosis: a study from the EULAR Scleroderma Trials and Research (EUSTAR) database. Ann Rheum Dis. 2010 Oct;69(10):1809-15. doi: 10.1136/ard.2009.114264. Epub 2010 Jun 15. PMID 20551155
- [Background] Hoyles RK, Ellis RW, Wellsbury J, Lees B, Newlands P, Goh NS, Roberts C, Desai S, Herrick AL, McHugh NJ, Foley NM, Pearson SB, Emery P, Veale DJ, Denton CP, Wells AU, Black CM, du Bois RM. A multicenter, prospective, randomized, double-blind, placebo-controlled trial of corticosteroids and intravenous cyclophosphamide followed by oral azathioprine for the treatment of pulmonary fibrosis in scleroderma. Arthritis Rheum. 2006 Dec;54(12):3962-70. doi: 10.1002/art.22204. PMID 17133610
- [Background] Keir GJ, Maher TM, Hansell DM, Denton CP, Ong VH, Singh S, Wells AU, Renzoni EA. Severe interstitial lung disease in connective tissue disease: rituximab as rescue therapy. Eur Respir J. 2012 Sep;40(3):641-8. doi: 10.1183/09031936.00163911. Epub 2012 Jan 26. PMID 22282550
- [Background] Goh NS, Desai SR, Veeraraghavan S, Hansell DM, Copley SJ, Maher TM, Corte TJ, Sander CR, Ratoff J, Devaraj A, Bozovic G, Denton CP, Black CM, du Bois RM, Wells AU. Interstitial lung disease in systemic sclerosis: a simple staging system. Am J Respir Crit Care Med. 2008 Jun 1;177(11):1248-54. doi: 10.1164/rccm.200706-877OC. Epub 2008 Mar 27. PMID 18369202
- [Derived] Maher TM, Tudor VA, Saunders P, Gibbons MA, Fletcher SV, Denton CP, Hoyles RK, Parfrey H, Renzoni EA, Kokosi M, Wells AU, Ashby D, Szigeti M, Molyneaux PL; RECITAL Investigators. Rituximab versus intravenous cyclophosphamide in patients with connective tissue disease-associated interstitial lung disease in the UK (RECITAL): a double-blind, double-dummy, randomised, controlled, phase 2b trial. Lancet Respir Med. 2023 Jan;11(1):45-54. doi: 10.1016/S2213-2600(22)00359-9. Epub 2022 Nov 11. PMID 36375479
- [Derived] Saunders P, Tsipouri V, Keir GJ, Ashby D, Flather MD, Parfrey H, Babalis D, Renzoni EA, Denton CP, Wells AU, Maher TM. Rituximab versus cyclophosphamide for the treatment of connective tissue disease-associated interstitial lung disease (RECITAL): study protocol for a randomised controlled trial. Trials. 2017 Jun 15;18(1):275. doi: 10.1186/s13063-017-2016-2. PMID 28619061